CLINICAL TRIAL: NCT04943666
Title: The Russian Multicenter Observational Study "Evaluation of the HDQ for the Diagnosis of Hemorrhoidal Disease ( HDQ )
Acronym: HDQ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05682-063-RUS
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Haemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hemorrhoid Disease Questionnaire — a new patient specific questionnaire (HDQ) with appropriate sensitivity and specificity to use for screening of patients with haemorrhoids in Russia in clinical practice for wider screening of haemorrhoids in population and for increasing patients' awareness of the disease and prompting them to seek professional advice.

SUMMARY:
Currently in Russia there is no available self-evaluating tools with appropriate diagnostic accuracy for screening of patients with haemorrhoids. Therefore, the primary objective of this study is to evaluate a new patient specific questionnaire (HDQ) with appropriate sensitivity and specificity to use for screening of patients with haemorrhoids in Russia. Once evaluated, the HDQ will be used in clinical practice for wider screening of haemorrhoids in population and for increasing patients' awareness of the disease and prompting them to seek professional advice.

Secondary objectives of the study are to describe a prevalence of haemorrhoids among patients in the study and to describe a prevalence of the symptoms of haemorrhoids among patients in the study

DETAILED DESCRIPTION:
Main parameters (primary outcomes) to be evaluated in the study are:

1. sensitivity of the HDQ for screening of patients with haemorrhoids;
2. specificity of the HDQ for screening of patients with haemorrhoids;

Additional parameters (secondary outcomes) in the study are:

1. Prevalence rate of haemorrhoids among study population established by physicians basing on the results of the objective examination;
2. Prevalence of the symptoms of haemorrhoids among patients in the study

ELIGIBILITY:
Inclusion Criteria:

* The patient came to visit a coloproctologist
* Male or female aged over 18 years
* Signed informed consent form to participate in the study has been obtained
* Absence of conditions requiring emergency medical care.
* The patient is not taking VAD for at least 1 month before the date on inclusion to the study

Exclusion Criteria:

* Confirmed or suspected malignant tumor
* Diagnosed coloproctological disease at the time of inclusion
* Severe somatic disorders (of heart and blood vessels, lungs, kidneys, pancreas, or liver), associated with decompensation of organ functions
* Mental disorders
* Presence of contraindications for examination

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: consecutive patients seeking help from a coloproctologist Limit: 450 characters.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity of the HDQ for screening of patients with haemorrhoids | 1 month
  Objective examination by physicians will be made that is required to determine the sensitivity of the patient's HDQ.
specificity of the HDQ for screening of patients with haemorrhoids; | 1 month
  Objective examination by physicians will be made that is required to determine the specificity of the patient's HDQ

SECONDARY OUTCOMES:
Prevalence rate of haemorrhoids among study population established by physicians basing on the results of the objective examination; | 1 month
  - to describe a prevalence of haemorrhoids among patients in the study
Prevalence of the symptoms of haemorrhoids among patients in the study | 1 month
  - to describe a prevalence of the symptoms of haemorrhoids among patients in the study

CONTACTS AND LOCATIONS:
Overall Officials: Yuriy Stoyko, Professor, Principal Investigator
Locations (1):
- National Medical and Surgical Center. N.I. Pirogov, Moscow, Russia